CLINICAL TRIAL: NCT02865070
Title: A Smart, "Always -On" Health Monitoring System, Sub-Study: No Strings Attached: Wireless Sensor Technology in the Prentice NICU
Brief Title: A Smart, "Always -On" Health Monitoring System
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Professor in Dermatology and Pediatrics, Northwestern University
Other Study IDs: MA06072012
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Premature Birth
Keywords: premature; wireless vitals; vitals monitor
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- 2 infants (ages 1-6mo) non-NICU setting
  Interventions: Device: Skin Sensor
- 10 babies (full term, ages 37-42 weeks)
  Interventions: Device: Skin Sensor
- 5 babies (premature, ages 34-37 weeks)
  Interventions: Device: Skin Sensor
- 5 babies (premature, ages 31-34 weeks)
  Interventions: Device: Skin Sensor
- 5 babies (premature, ages 28-31 weeks)
  Interventions: Device: Skin Sensor
- 5 babies (premature, ages 25-28 weeks)
  Interventions: Device: Skin Sensor
- 5 babies (premature, ages 23-25 weeks)
  Interventions: Device: Skin Sensor
- 30 babies (any gestational age under 6 months)
  Interventions: Device: Skin Sensor
- 25 neonates (ages 24-29 weeks for sub-study)
  Interventions: Device: Skin Sensor

INTERVENTIONS:
Device: Skin Sensor — Wireless vitals monitor

SUMMARY:
This is a pilot study is to test a wireless, skin-sensor device against current technology in the NICU to monitor vitals

DETAILED DESCRIPTION:
This is a single center, prospective, observational study that will recruit subjects from Lurie Children's Hospital and Prentice Women's Hospital to test a new wireless vitals monitor against the current vitals monitors used in the NICU. Patients will be neonates in different age brackets.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in different age cohorts from ages 25 weeks gestational age to fullterm infants or infants up to 6 months of age, selected with assistance of NICU staff
* Currently in NICU and requiring monitoring for heart rate, ECG, respiratory rate, temperature, and pulse oximetry
* Parents able to understand and provide informed consent for study
* Infants enrolled in the Pre-Vent study (sub-study only)

Exclusion Criteria:

* Over 6 months of age
* Hemodynamic or other instability precluding testing of new monitoring with concurrent standards
* Infants at imminent risk of death and neonates with a skin abnormality that precludes assessment

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 110 premature babies in the Lurie Children's Hospital and Prentice Women's Hospital NICU within 1 week of birth that fall into one of the listed cohorts, fit inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Correlation of vital parameters against current technology | 15 min, 3 hours, 24 hours, 1 week

SECONDARY OUTCOMES:
Adverse events from wireless monitoring sensor assessed through Neonatal Skin Condition Score (NSCS)-sub-study only | 24 hours, 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University, Lurie Children's Hospital Department of Dermatology
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States